CLINICAL TRIAL: NCT00688064
Title: Efficacy and Safety Comparison of Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel Associated With Doxycycline Hyclate 100 mg Tablets Versus Adapalene 0.1% / Benzoyl Peroxide 2.5% Vehicle Gel Associated With Doxycycline Hyclate 100 mg Tablets in the Treatment of Severe Acne Vulgaris.
Brief Title: Adapalene-BPO Gel Associated With Doxycycline Hyclate 100 mg in the Treatment of Severe Acne Vulgaris
Acronym: ACCESS I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Jean-Charles DHUIN Clinical Trial Manager, Galderma
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.03.SPR.29074
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Results first posted 2010-03-31 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2010-03

CONDITIONS: Severe Acne Vulgaris
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Adapalene-BPO + Doxycyline
  Interventions: Drug: Adapalene BPO Gel associated with Doxycyline Hyclate
- 2 (Active Comparator): Vehicle + Doxycycline
  Interventions: Drug: Vehicle Gel associated with Doxycycline Hyclate

INTERVENTIONS:
Drug: Adapalene BPO Gel associated with Doxycyline Hyclate — Adapalene BPO Gel: Topical to the face, once daily in the evening Doxycycline Hyclate: Oral, 1 tablet once daily in the morning. Both during 12 weeks.
  Other Names: Adapalene-BPO gel + Doxycycline
  Arms: 1
Drug: Vehicle Gel associated with Doxycycline Hyclate — Vehicle Gel: Topical to the face, once daily in the evening; Doxycycline Hyclate: Oral, 1 tablet once daily in the morning. Both during 12 weeks.
  Other Names: Vehicle gel + Doxycycline
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the efficacy of Adapalene 0.1% / Benzoyl Peroxide (quoted as BPO) 2.5% Gel associated with Doxycycline Hyclate 100 mg Tablets compared to Adapalene 0.1% /Benzoyl Peroxide 2.5% Vehicle Gel associated with Doxycycline Hyclate 100 mg Tablets, in the treatment of severe acne vulgaris. The safety of the two treatment regimens will also be evaluated.

DETAILED DESCRIPTION:
Further to this study, eligible Subjects with at least good Global Assessment of Improvement at Week 12 will be randomized in a maintenance study (SPR.29075)

ELIGIBILITY:
Inclusion Criteria:

* Male or female Subjects of any race, aged 12 to 35 years inclusive
* Subjects with severe facial acne (global severity score of 4)
* Subjects with a minimum of 20 inflammatory lesions (papules and pustules) on the face, excluding the nose
* Subjects with a minimum of 30 and a maximum of 120 non-inflammatory lesions (open comedones and closed comedones) on the face, excluding the nose

Exclusion Criteria:

* Subjects with more than 3 nodules or cysts on the face,
* Subjects with acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc.)

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 459 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Stein Gold, MD, Principal Investigator — Henry Ford Medical Center-New Center One, Detroit, MI
Locations (34):
- United States (28):
  - Galderma Investigational Site, Oceanside, California
  - Galderma Investigational Site, San Diego, California
  - Galderma Investigational Site, Denver, Colorado
  - Galderma Investigational Site, Longmont, Colorado
  - Galderma Investigational Site, Miami, Florida
  - Galderma Investigational Site, Snellville, Georgia
  - Galderma Investigational Site, Chicago, Illinois
  - Galderma Investigational Site, Evansville, Indiana
  - Galderma Investigational Site, Overland Park, Kansas
  - Galderma Investigational Site, Louisville, Kentucky
  - Galderma Investigational Site, Detroit, Michigan
  - Galderma Investigational Site, Fort Gratiot, Michigan
  - Galderma Investigational Site, Fridley, Minnesota
  - Galderma Investigational Site, Omaha, Nebraska
  - Galderma Investigational Site, Albuquerque, New Mexico
  - Galderma Investigational Site, Stony Brook, New York
  - Galderma Investigational Site, Winston-Salem, North Carolina
  - Galderma Investigational Site, Warren, Ohio
  - Galderma Investigational Site, Hazleton, Pennsylvania
  - Galderma Investigational Site, Hershey, Pennsylvania
  - Galderma Investigational Site, Simpsonville, South Carolina
  - Galderma Investigational Site, Arlington, Texas
  - Galderma Investigational Site, Austin, Texas
  - Galderma Investigational Site, College Station, Texas
  - Galderma Investigational Site, Houston, Texas
  - Galderma Investigational Site, Lubbock, Texas
  - Galderma Investigational Site, San Antonio, Texas
  - Galderma Investigational Site, Webster, Texas
- Canada (4):
  - Galderma Investigational Site, Barrie, Ontario
  - Galderma Investigational Site, North Bay, Ontario
  - Galderma Investigational Site, Windsor, Ontario
  - Galderma Investigational Site, Québec, Quebec
- Puerto Rico (2):
  - Galderma Investigational Site, Aibonito
  - Galderma Investigational Site, Carolina

REFERENCES:
- See also: Related Info — http://www.galderma.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 18 AUG 2008 to 14 NOV 2008 in thirty-five centers (30 in the USA and 5 in Canada) public or private practices. Twenty-five USA centers and four Candadian centers used a central IRB, and the others used a local IRB.
Groups:
- Adapalene-BPO + Doxycycline: Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel associated with Doxycyline Hyclate 100 mg tablet.
- Vehicle + Doxycycline: Vehicle Gel associated with Doxycycline Hyclate 100 mg tablet
Period: Overall Study
Arm/Group | Adapalene-BPO + Doxycycline | Vehicle + Doxycycline
Started | 232 | 227
Completed | 211 | 201
Not Completed | 21 | 26
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 2 | 4
Not completed — Withdrawal by Subject | 7 | 7
Not completed — Lost to Follow-up | 10 | 10
Not completed — Lack of Efficacy | 0 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Any other reasons | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adapalene-BPO + Doxycycline | Vehicle + Doxycycline | Total
Number analyzed (Participants) | 232 | 227 | 459
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 152 | 156 | 308
  Between 18 and 65 years | 80 | 71 | 151
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.6 (5.84) | 18.1 (4.92) | 18.4 (5.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 97 | 205
  Male | 124 | 130 | 254
Region of Enrollment [Number; unit: participants]
  United States | 170 | 164 | 334
  Puerto Rico | 18 | 18 | 36
  Canada | 44 | 45 | 89

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Total Lesion Counts at Week 12.
Time Frame: Week 12
Population: ITT, LOCF
Measure: Median (Full Range); unit: % of change
Arm/Group | Adapalene-BPO + Doxycycline | Vehicle + Doxycycline
Number analyzed (Participants) | 232 | 227
% of change | -64 [-100 to 34] | -41 [-92 to 64]

2. Secondary Outcome: Percent Change From Baseline in Inflammatory Lesion Counts at Week 12.
Time Frame: Week 12
Population: ITT, LOCF
Measure: Median (Full Range); unit: % of change
Arm/Group | Adapalene-BPO + Doxycycline | Vehicle + Doxycycline
Number analyzed (Participants) | 232 | 227
% of change | -72 [-100 to 59] | -48 [-93 to 79]

3. Secondary Outcome: Percent Change From Baseline in Non-inflammatory Lesion Counts at Week 12
Time Frame: Week 12
Population: ITT, LOCF
Measure: Median (Full Range); unit: % of change
Arm/Group | Adapalene-BPO + Doxycycline | Vehicle + Doxycycline
Number analyzed (Participants) | 232 | 227
% of change | -61 [-100 to 81] | -40 [-98 to 149]

4. Secondary Outcome: Success Rate on the Investigator's Global Assessment
Description: Percentage of subjects graded "Clear" or "Almost Clear" on 6-point IGA scale(0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe and 5=very severe)at week 12
Time Frame: Week 12
Population: ITT, LOCF
Measure: Number; unit: % of subjects
Arm/Group | Adapalene-BPO + Doxycycline | Vehicle + Doxycycline
Number analyzed (Participants) | 232 | 227
% of subjects | 31.5 | 8.4

5. Secondary Outcome: Percent of Subjects With Adverse Events
Description: Percent of subjects with Adverse Events all along the study (up to 12 weeks follow-up period)
Time Frame: Up to 12 weeks
Population: ITT
Measure: Number; unit: % of subjects
Arm/Group | Adapalene-BPO + Doxycycline | Vehicle + Doxycycline
Number analyzed (Participants) | 232 | 227
% of subjects | 26.3 | 26.9

ADVERSE EVENTS:
Arm/Group | Adapalene-BPO + Doxycycline | Vehicle + Doxycycline
Serious Adverse Events (participants affected / at risk) | 0/232 | 0/227
Other Adverse Events (participants affected / at risk) | 43/232 | 48/227
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapalene-BPO + Doxycycline (N=232) | Vehicle + Doxycycline (N=227)
dyspepsia (Gastrointestinal disorders) | 2 (2) | 5 (5)
gastroenteritis viral (Infections and infestations) | 5 (5) | 2 (2)
nasopharyngitis (Infections and infestations) | 10 (10) | 13 (14)
nausea (Gastrointestinal disorders) | 9 (9) | 12 (14)
upper respiratory tract infection (Infections and infestations) | 8 (8) | 6 (6)
vomiting (Gastrointestinal disorders) | 9 (10) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any intent of the investigator to publish or disclose in any way the information requires the sponsor's prior written approval. The investigator shall provide their draft of such publication to sponsor for review and approval at least 2 months prior to the date of the intended publication. Sponsor shall have the absolute right to determine whether information may be published by the investigator.